CLINICAL TRIAL: NCT00498537
Title: Spironolactone for Reducing Proteinuria in Diabetic Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Saklayen, Mohammad - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0024
Record Dates: First submitted 2007-07-06; First posted 2007-07-10 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-05

CONDITIONS: Diabetic Nephropathy
Keywords: spironolactone; aldosterone; diabetic nephropathy; proteinuria; hyperkalemia; albuminuria; renal failure
MeSH Terms: conditions — Diabetic Nephropathies; Proteinuria; Hyperkalemia; Albuminuria; Renal Insufficiency | interventions — Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other)
  Interventions: Drug: spironolactone
- 2 (Other)
  Interventions: Drug: spironolactone

INTERVENTIONS:
Drug: spironolactone

SUMMARY:
Introduction: Aldosterone seems to have deleterious effects on the kidneys. Many animal studies and few clinical trials now have shown that suppression of aldosterone by aldosterone receptor blockers ameliorated these effects.

Method: In a double-blind, cross over study, 24 patients with diabetic nephropathy who were already receiving either ACE inhibitor(lisinopril 20-40 mg/day ) or ARB( losartan 25-100 mg/day )were given spironolactone( 25 mg during the first month and 50 mg during the second and third month if serum K remained ok) or matching placebo with 1 month of washout in between. All patients were from a single center and exclusively male veterans. Blood pressure, serum creatinine, serum K and spot urine protein/creatinine were measured at the beginning and end of each study period. The study was started in May of 2003 and completed in May 2006.

DETAILED DESCRIPTION:
Spironolactone for reducing proteinuria and progression of renal failure in diabetic nephropathy

Introduction:

Diabetic nephropathy is the leading cause of ESRD in USA now and accounts for 40% of all new patients that begins renal replacement therapy each year. The number of new patients starting chronic dialysis therapy is 70,000 each year and is increasing. This number does not include patients who decline dialysis therapy or die soon after starting dialysis. The economic and human cost of diabetic nephropathy is therefore enormous.

Aggressive control of blood pressure especially with ACE-inhibitor had been shown to reduce proteinuria and progression of renal dysfunction in both type 1 and type 2 diabetics. Use of ACE-inhibitor reduced proteinuria even in normotensive diabetics with microalbuminuria. However even with optimal use of ACE-Inhibitor the progression of renal dysfunction is not completely stopped. Other additional treatment strategies therefore need to be explored.

Studies in animals and small pilot studies in humans have shown that nondihydropyridine calcium channel blockers (e.g. diltiazem or verapamil) may have additional protective effect in reducing proteinuria when used in conjunction with ACE-inhibitor. Use of angiotensin receptor blockers along with ACE-inhibitors also had been tried but results are not dependable because of the short sample size.

While angiotensin plays the major role in glomerular hemodynamics there is increasing evidence that aldosterone plays a significant role in renal hemodynamics independent of angiotensin. In a remnant kidney model in the rat Greene et al showed that there was greater than 10-fold rise in aldosterone in the remnant kidney rats (REM) compared to SHAM operated ones. As expected, the proteinuria, hypertension and glomerulosclerosis in the REM rats were attenuated with treatment with ACE-inhibitor and angiotensin receptor blockers (REM AIIA). However when these rats (REM AIIA) were treated with aldosterone infusion the proteinuria, hypertension and glomerulosclerosis seen were similar to REM alone rats, suggesting deleterious renal hemodynamic effects of aldosterone independent of angiotensin II. Use of spironolactone in these rats transiently reduced proteinuria and lowered arterial pressure.

Previous experiment in remnant kidney model also showed that adrenalectomy with adequate glucocorticoid replacement reduced the proteinuria and other evidence of renal injury usually seen in REM rats. Similarly heparin administration provides remarkably complete protection from injury in remnant kidney model. Although this effect could be due to any of several actions of heparin (anticoagulant and hemodynamic), it could be due to known suppressive action of heparin on aldosterone synthesis.

In stroke-prone spontaneously hypertensive rats (SHRSP), renal vascular injury causing proteinuria and malignant nephrosclerotic lesions were markedly reduced by treatment with spironolactone, an aldosterone receptor blocker. The effect of spironolactone alone was comparable to effect of treatment with captopril, an ACE-inhibitor. In further studies Rocha et al had shown that the ameliorating effect of ACE-inhibition in the SHRSP rats could be fully reversed by infusion of aldosterone, suggesting a major role for aldosterone in the vascular injury in these rats as well. Importantly the deleterious effect of aldosterone and the protective effect of spironolactone against end organ damage in SHRSP rats appeared to be independent of the blood pressure effects.

In another experiment, the Wistar-Furth rat, an inbred strain resistant to actions of mineralocorticoids, was used to study the concept that mineralocorticoids contribute to progressive renal injury. Renal damage, as evidenced by albuminuria and glomerulosclerosis, in response to 5/6 nephrectomy was markedly less in Wistar-Furth rats compared to Wistar rats. Treatment of hypertension seen in the nephrectomized Wistar rats did not protect them from renal injury suggesting again that mineralocorticoid mediated deleterious effect was independent of the blood pressure effect.

Hyperaldosteronism has been noted as a component of clinical chronic renal insufficiency of various etiologies. In a cross sectional study of patients with mild to moderate renal insufficiency Hene et al observed that level of serum aldosterone increased as creatinine clearance fell below 70 cc/min and went up as high as 3-4 fold the baseline. Similarly in a study of 9 patients with average inulin clearance of 27cc/min, Bauer and Reams noted plasma aldosterone level to be four fold greater than normal. The significance of this Hyperaldosteronism as to the progression of the renal insufficiency had not been studied systematically, but in one longitudinal study Walker noted a significant correlation between aldosterone level and rate of progression of renal failure. In this longitudinal study of 131 diabetic cohort, Walker noted that hypertension, plasma angiotensin II and aldosterone were independent predictors of accelerated loss of renal function.

Although the distal tubule is considered the target for aldosterone action, aldosterone receptors had been found in myocardium, vascular smooth muscle cells and glomeruli .In vitro studies of cultured mesangial cells revealed increased production of type IV collagen after incubation with aldosterone. In a double blind controlled study MacFadyen and colleagues observed that spironolactone treatment reduced circulating levels of procollagen type III N-terminal amino peptide, a marker of vascular collagen turnover. Weber and other investigators have observed that aldosterone caused myocardial fibrosis and this effect could be ameliorated by treatment with spironolactone. In addition to the classical genomic action through the type 1 mineralocorticoid receptor, aldosterone is now known to have significant non-genomic mediated action in many different tissues including kidney tubules and vascular smooth muscle cells. Aldosterone also up regulates Angiotensin II membrane receptors thereby multiplying the vascular effect of Ang II. This upregulation was inhibited by treatment with spironolactone. These findings are consistent with a synergistic action between Ang II and aldosterone in the production of vascular injury as first proposed by Masson et al almost 4 decades ago.

The use of ACE inhibitors may strongly inhibit the RAAS, but their suppressive effect on aldosterone production may not be satisfactory. Indeed, in hypertension as well as in CHF, continuous treatment with ACE inhibitor did not produce a sufficient decrease in plasma aldosterone level, which remained high or increases eventually during long term use. In one study, patients treated with hefty doses of captopril (300 mg/day) had a doubling of the plasma aldosterone level at the end of 12 months of therapy despite marked decrease in ANG II level. The reasons for the unsatisfactory suppressive effect of ACE inhibitors on plasma aldosterone could be partly due to tachyphylaxis and also very likely due to predominance of the non-RAAS component of the control system for aldosterone production. Urinary clearance of aldosterone may also be reduced in CHF and CRF. On the basis of these understandings, spironolactone (25-50 mg a day) was used in a large multi-centered randomized controlled trial for treatment of congestive heart failure who already were receiving standard therapy with Ace inhibitors, diuretics and digoxin. The study was terminated in midway because interim analysis showed 30% reduction in mortality in the spironolactone treated group as opposed to the control. Of note, the incidence of hyperkalemia in the treatment group was only 1.7% as opposed to 1% in the placebo group. The incidence of gynecomastia was also modest (10% Vs 1%) in spite of use of other drugs like digoxin that are known also to cause gynecomastia.

Planned Study:

For this study we will recruit patients from the renal clinic at the VA medical center and also some patients from the primary care clinics at the same hospital. The study will be a double blind control study using each patient as his own control after a period of wash out phase.

Inclusion criteria

Patients with diabetic nephropathy (with proteinuria exceeding 100 mg per day while on ace inhibitor ) who are already being treated with ACE-Inhibitor at maximum tolerated dose. For lisinopril this dose usually will be 20-40 mg per day. Patients who are on angiotensin receptor blocker ( ARB ) due to inability to tolerate ace inhibitor ( e.g. due to cough ) will be also considered for the study provided they stay on the same ARB at same dose throughout the study period.

Exclusion criteria:

Serum creatinine greater than 2.0 mg/dl Serum K greater than 5.0 meq/L Patients who need to use spironolactone for some other reasons Life expectancy less than 1 year For this pilot phase of the study we will investigate 30 patients (see attached sample size calculation) equally divided into control and treatment groups. Patients will be randomly allocated to the different groups by using computer generated randomization sequence. After 3 months on study medication (or placebo) the study group of patients will be switched to the placebo group and vice versa. Thus each patient will be his own control. There will be a month of wash out period in between this change over.

Study drug:

Study drug will be spironolactone. The starting dose will be 25 mg orally every day, which will be increased to 50 mg every day, if tolerated after 4 weeks. A matching placebo will be used for the placebo group. The VA pharmacy will prepare and provide the study drug as well as the placebo. The pharmacy will create and maintain the randomization numbers in a safe place so that the investigators and the study nurses remain blind to the whole randomization process all throughout the study period.

Protocol of lab studies and follow up:

All patients will be seen by one of the investigator and have a brief history and physical examination prior to randomization. All patients will have their blood pressured measured by a study nurse in a sitting position (average of two BP readings taken at 5 minutes interval will be recorded). Patients will be weighed at each visit also.

The study related visits would be prior to randomization, day of randomization, at 1 month and at 3 month in study.

The cycle will be repeated again for each patient after one month washout period after which their study drug will be reversed (placebo to study and study to placebo)

All patients will have the following lab studies at the beginning (prior to randomization), at 1 month and at 3 month clinic visits:

Renal panel 24 hours urine for protein and creatinine Renal panel can be done in between the prescribed study visits for clinical reasons.

All patients will be continued on their other usual medication during the study period and changes will be made as deemed necessary by the clinicians taking care of patients. As far as possible the dose of ace inhibitor (or angiotensin receptor blocker) will be kept the same as at the beginning of randomization. Doses of calcium channel blocker (if they are on it) will also not be changed as much as possible during the study.

ELIGIBILITY:
Inclusion Criteria:

The study is completed. Inclusion criteria was diabetic nephropathy

Exclusion Criteria:

Scr >2 mg/dl and serum K > 5meq/L

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-01; Primary Completion 2005-12 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
reduction in proteinuria

SECONDARY OUTCOMES:
Changes in GFR and incidence of hyperkalemia

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad G. Saklayen, MD, Principal Investigator — VA Medical Center, Dayton
Locations (1):
- VA Medical Center, Dayton, Dayton, Ohio, United States

REFERENCES:
- [Result] Saklayen MG, Gyebi LK, Tasosa J, Yap J. Effects of additive therapy with spironolactone on proteinuria in diabetic patients already on ACE inhibitor or ARB therapy: results of a randomized, placebo-controlled, double-blind, crossover trial. J Investig Med. 2008 Apr;56(4):714-9. doi: 10.2310/JIM.0b013e31816d78e9. PMID 18382267
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592